CLINICAL TRIAL: NCT00080002
Title: Effectiveness and Safety Study of Pegamotecan (PEG-Camptothecin) in Patients With Locally Advanced or Metastatic Cancer of the Stomach or Gastroesophageal Junction Who Have Relapsed or Progressed Following a Previous Chemotherapy Treatment
Brief Title: Efficacy of Pegamotecan (PEG-Camptothecin) in Localized or Metastatic Cancer of the Stomach or Gastroesophageal Junction
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Enzon Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAM-9011
Record Dates: First submitted 2004-03-19; First posted 2004-03-23 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2005-03

CONDITIONS: Cancer of Stomach; Gastroesophageal Cancer
Keywords: cancer; gastric; gastroesophageal junction; neoplasms; gastric cancer; gastric neoplasms
MeSH Terms: conditions — Stomach Neoplasms; Neoplasms | interventions — pegamotecan

INTERVENTIONS:
Drug: Pegamotecan

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of pegamotecan (PEG-camptothecin) in patients with pathologically-diagnosed locally advanced or metastatic adenocarcinoma of the stomach or gastroesophageal junction who have relapsed or progressed following one prior chemotherapy treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of adenocarcinoma of the stomach or gastroesophageal junction.
* Disease measurable in at least one dimension.
* Target tumors outside of prior radiation field(s).
* An Eastern Cooperative Oncology Group (ECOG) performance scale score of 0 or 1
* Adequate hematologic profile, as determined by hemoglobin, platelet, and neutrophil count.
* Adequate renal function, as determined by serum creatinine and serum albumin measurements.
* Adequate liver function, as determined by total bilirubin and transaminases levels. Transaminases may be <= 5.0x ULN if due to metastatic disease in the liver.
* Fully recovered from prior surgery.
* No history of hemorrhagic cystitis.
* No microscopic hematuria (>10 RBC/hpf) unless documented to be due to an infection or non-bladder origin.
* Capable of understanding the protocol requirements and risks and providing written informed consent.

Exclusion Criteria:

* Concurrent serious medical illness unrelated to tumor within the past 6 months.
* Known chronic infectious disease, such as AIDS or hepatitis (screening for hepatitis and HIV will not be performed).
* Positive screening pregnancy test or is breast-feeding.
* Female or male subject of reproductive capacity who is unwilling to use methods appropriate to prevent pregnancy during the course of this study.
* Receiving concurrent chemotherapy, investigational agents, radiotherapy, surgery, or has received wide field radiation within the previous 4 weeks.
* History of another malignancy (except basal and squamous cell carcinomas of the skin and carcinoma in situ of the cervix) within the last 5 years.
* Known or clinically suspected brain metastases.
* Received more than one prior regimen of chemotherapy for locally advanced or metastatic adenocarcinoma of the stomach or GE junction.
* Received prior neoadjuvant and/or adjuvant cytotoxic chemotherapy
* Received any investigational drug within the last 30 days.
* Not fully recovered from any prior, and from any reversible side effects related to the administration of cytotoxic chemotherapy, investigational agents, or radiation therapy.
* Prior treatment with a camptothecin analog.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-12